CLINICAL TRIAL: NCT02918929
Title: A Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study of Orally Administered EDP-305 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (SAD), Multiple Ascending Doses (MAD) and the Effect of Food on EDP-305 Pharmacokinetics in Healthy Subjects, and of Multiple Ascending Doses (MAD) in Subjects With Presumptive NAFLD
Brief Title: A Study of EDP 305 in Healthy Subjects and Subjects With Presumptive NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 305-001
Record Dates: First submitted 2016-08-29; First posted 2016-09-29 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Presumptive NAFLD
Keywords: First-in-human; Single Ascending Dose; Multiple Ascending Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- EDP 305 SAD Cohorts (Experimental): EDP 305 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5, and Dose 6 oral suspension, once daily in one single administration
  Interventions: Drug: EDP 305
- EDP 305 MAD Cohorts (Experimental): EDP 305 Dose 1, Dose 2, Dose 3, Dose 4, Dose 5 and Dose 6 oral suspension, once daily for 14 days
  Interventions: Drug: EDP 305
- EDP 305 SAD Placebo Cohort (Placebo Comparator): Matching placebo, oral suspension, once daily in one single administration
  Interventions: Drug: Placebo
- EDP 305 MAD Placebo Cohort (Placebo Comparator): Matching placebo, oral suspension, once daily for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP 305
  Arms: EDP 305 MAD Cohorts; EDP 305 SAD Cohorts
Drug: Placebo — placebo to match EDP 305
  Arms: EDP 305 MAD Placebo Cohort; EDP 305 SAD Placebo Cohort

SUMMARY:
This randomized, double-blind, placebo-controlled study will assess the safety, tolerability, and pharmacokinetics of single and multiple orally administered doses of EDP-305 in healthy adult subjects, and adult subjects with presumptive NAFLD (i.e., obese subjects with or without prediabetes or T2DM).

DETAILED DESCRIPTION:
The first phase assesses single ascending doses for EDP 305 (active drug or placebo) in healthy subjects. A "fasted" and "fed" two-part cohort will also assess food effect.

The second phase assesses multiple ascending doses (active drug or placebo) for 14-days in healthy subjects and also in subjects with presumptive NAFLD (i.e., obese subjects with or without prediabetes or T2DM).

Each cohort within each phase will enroll a total of 8 subjects who will be randomized to receive EDP-305 or placebo. The cohort assessing food effect will enroll 10 subjects randomized to receive EDP-305 or placebo.

ELIGIBILITY:
Inclusion Criteria for all SAD and MAD Subjects::

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Female subjects must be of non-childbearing potential.
* All male participants who have not had a vasectomy must use effective contraception from Day -1 to 90 days after their last dose of study drug.
* For healthy volunteers only (see below for Subjects with presumptive NAFLD): Body mass index of 18 to 30 kg/m2 with a minimum body weight of 50 kg.

Additional Inclusion Criteria for MAD Subjects with Presumptive NAFLD:

* Body mass index of >28 and <35 kg/m2 at screening.

WITH or WITHOUT one of the following:

* Type 2 diabetes mellitus diagnosed by one of the following methods:

  * As defined by the American Diabetes Association (ADA), as one of the following criteria: a) symptoms of diabetes plus casual plasma glucose concentration >200 mg/dL (11.1 mmol/L) OR b) Fasting plasma glucose >126 mg/dL (7.0 mmol/L) OR c) 2-hour post-load glucose >200 mg/dL (11.1 mmol/L) during a 75 g oGTT.
  * HbA1c of at least 6.5%. --- OR---
* Prediabetes diagnosed as defined by the ADA as a) an HbA1c of 5.7% - 6.4% OR b) fasting blood glucose of 100-125 mg/dL OR c) an oGTT 2-hour blood glucose of 140 mg/dL - 199 mg/dL.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption
* Participation in a clinical trial within 30 days prior to study drug administration.
* Use of prescription drugs, non-prescription drugs, dietary supplements including Vitamin E herbal supplements, hormonal therapy/replacement or CYP3A4 substrates, inducers and inhibitors within 14 days prior to the first dose of study medication.

Additional Exclusion Criteria for MAD Subjects with Presumptive NAFLD:

* Subjects taking any antidiabetic medication.
* Subjects with unstable proliferative retinopathy, macular oedema (fundus examination performed in the previous year will be considered relevant on Investigator's judgement).
* Subject has taken fibrates, statins, and/or Vitamin E within 6 weeks prior to the first dose administration.
* Subjects with a history of bariatric surgery and any other gastrointestinal surgery relative to weight loss.
* Subjects with common causes of secondary hepatic steatosis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety data including but not limited to adverse events, physical exams, vital signs, 12-lead ECGs and clinical lab results (including chemistry, hematology, and urinalysis). | From screening to the 7-day post treatment safety follow up visit.

SECONDARY OUTCOMES:
Cmax | 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72 (D4), and 96 (D5) hrs post dose.
  EDP 305
Cmax | Day 1: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15 hrs; Days 2, 3, 4, 5, 7, 9, 12; Day 14: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24 (D15), 30, 36, 48 (D16), 60, 72 (D17), and 96 (D18) hrs postdose
  EDP 305
AUC | 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24, 30, 36, 48, 60, 72 (D4), and 96 (D5) hrs post dose.
  EDP 305
AUC | Day 1: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15 hrs; Days 2, 3, 4, 5, 7, 9, 12; Day 14: 0 (predose), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 24 (D15), 30, 36, 48 (D16), 60, 72 (D17), and 96 (D18) hrs postdose
  EDP 305

OTHER OUTCOMES:
Change from baseline: FGF19 | Day 1 predose and postdose hours 2, 4, 8, 12, and 24 (i.e., Day 2 predose)
Change from baseline: C4 | Day 1 predose and postdose hours 2, 4, 8, 12, and 24 (i.e., Day 2 predose)
Change from baseline: FGF19 | Day 1 predose and postdose hours 2, 4, 6, 8, 12 and 24 (i.e., Day 2 predose); Day 7 predose and postdose hours 8, 12, and 24 (i.e., Day 8 predose); Day 14 predose and postdose hours 8, 12, and 24 (i.e., Day 15 predose)
Change from baseline: C4 | Day 1 predose and postdose hours 2, 4, 6, 8, 12 and 24 (i.e., Day 2 predose); Day 7 predose and postdose hours 8, 12, and 24 (i.e., Day 8 predose); Day 14 predose and postdose hours 8, 12, and 24 (i.e., Day 15 predose)
Change from baseline: total bile acids | Day 1 predose and approximately 8 to 12 hours postdose
Change from baseline: total bile acids | Day 1 predose; Day 7 approximately 8 to 12 hours postdose; Day 14 approximately 8 to 12 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, MD, Principal Investigator — Pharmaceutical Research Associates
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
When the clinical study report has been submitted to the appropriate Regulatory authorities, a lay person summary will be provided to all study subjects by mail or email.